CLINICAL TRIAL: NCT00207155
Title: An Exploratory Pharmacogenomic Study of Monotherapy Erbitux in Subjects With Metastic Colorectal Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CA225-045
Record Dates: First submitted 2005-09-12; First posted 2005-09-21 (Estimated); Last update posted 2015-10-28 (Estimated); Status verified 2015-10

CONDITIONS: Metastatic Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Cetuximab

ARMS (1):
- A (Experimental)
  Interventions: Drug: Cetuximab

INTERVENTIONS:
Drug: Cetuximab — IV solution, IV, 400 mg/m2 initial dose + 250-400 mg/m2 weekly, Weekly, Until disease progression.
  Other Names: Erbitux

SUMMARY:
The purpose of this study is to predict response to Erbitux as a single agent in patients with metastatic colon cancer

ELIGIBILITY:
Inclusion Criteria:

* Measurable disease Tumor available for biopsies. Life expectancy of at least 3 months.

Exclusion Criteria:

* Known or documented brain metastases prior to Cetuximab therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110
Dates: Start 2003-12; Primary Completion 2006-02 (Actual); Study Completion 2006-02 (Actual)

PRIMARY OUTCOMES:
Prediction of response to Erbitux in subjects with metastatic colorectal cancer

SECONDARY OUTCOMES:
Radiographic Response

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (14):
- United States (12):
  - Local Institution, Duarte, California
  - Local Institution, Tampa, Florida
  - Local Institution, Baltimore, Maryland
  - Local Institution, St Louis, Missouri
  - Local Institution, New Brunswick, New Jersey
  - Local Institution, The Bronx, New York
  - Local Institution, Cincinnati, Ohio
  - Local Institution, Cleveland, Ohio
  - Local Institution, Hershey, Pennsylvania
  - Local Institution, Philadelphia, Pennsylvania
  - Local Institution, Nashville, Tennessee
  - Local Institution, San Antonio, Texas
- Local Institution, Montreal, Quebec, Canada
- Local Institution, Barcelona, Spain